CLINICAL TRIAL: NCT01432366
Title: Subcutaneous Anti-tnf-αlpha In Rheumatoid Arthritis: Analyze The Correlation Between Objective Measures Of Disease Activity And Safety And A Subjective Measure Such As Patient Beliefs About A Medicine
Brief Title: Correlation Between Beliefs About Medicine and Objective Measures of Efficacy and Safety in Rheumatoid Arthritis (RA)
Acronym: CONTENT
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-4746; B1801047 (Other: Alias Study Number)
Record Dates: First submitted 2011-08-18; First posted 2011-09-13 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients treated with SC anti-TNF
  Interventions: Other: SC anti-TNF

INTERVENTIONS:
Other: SC anti-TNF — Subcutaneous (SC) anti-TNF

SUMMARY:
It can be assumed that there is a link between what the patient feels and thinks about his medication and objective measures of disease activity and safety.

DETAILED DESCRIPTION:
A total of 500 subjects will provide 80% power to test the hypothesis that the absolute value of the correlation between two measures (e.g., BMQ Necessity and DAS28) is ≤ 0.3 (i.e., H0:│r│ ≤ 0.3 ) versus the alternative that it is > 0.3 (i.e., H1:│r │ > 0.3 ) assuming the absolute value of the true correlation is 0.40. A total of 500 will be enrolled to allow for approximately 5% being lost from analysis due to lack of post baseline data.

The Pearson method will be used for correlation between the BMQ total score for Necessity and the DAS28 and between the BMQ total score for Concern and DAS28. The Spearman rank method will be used for correlation between the BMQ total scores and Safety. For these latter analyses, subjects will be classified into one of 3 safety categories: (1) No AEs, (2) Non-serious AEs, (3) Serious AEs. 95% confidence intervals for the correlations will be provided.

ELIGIBILITY:
Inclusion Criteria:

Patients with RA on stable therapy defined as:

Etanercept: 1x50 mg/week or 2x25mg/week for at least 1 consecutive year. Adalimumab: 1x40 mg every other week for at least 1 consecutive year. Oral corticosteroids: stable doses for ≥ 12 weeks before baseline Methotrexate: stable doses for ≥ 12 weeks before baseline Other DMARD's: stable doses for ≥ 12 weeks before baseline

Exclusion Criteria:

Participation in other clinical or observational trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rheumatoid arthritis patients treated with SC anti-TNF capable of completing some questionnaires
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Algemeen Ziekenhuis St Jan, Bruges, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4746&StudyName=Correlation%20Between%20Beliefs%20About%20Medicine%20and%20Objective%20Measures%20of%20Efficacy%20and%20Safety%20in%20Rheumatoid%20Arthritis%20%28RA%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha): Participants with rheumatoid arthritis (RA), who were on stable therapy and received subcutaneous anti-TNF-alpha treatment for at least 1 consecutive year as per treating physician's discretion based on summary of product characteristics, were followed up for 1 year.
Period: Overall Study
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Started | 460
Completed | 392
Not Completed | 68
Not completed — Non-Responder | 7
Not completed — Adverse Event | 8
Not completed — Withdrawal Due to Non-Compliance | 3
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 13
Not completed — Lack of Efficacy | 1
Not completed — Site Closed | 20
Not completed — Investigator Forget to Complete Visits | 1
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Population: Baseline analysis set (BAS) included all participants who were enrolled in the study and seen at baseline.
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336
  Male | 124

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Beliefs About Medicines Questionnaire (BMQ) Necessity Score and Disease Activity Score Based on 28 Joints Count (DAS28) at Month 12
Description: Correlation between BMQ necessity and DAS28 was assessed by using Pearson correlation coefficient. BMQ necessity: 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicate degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). DAS28: calculated from number of swollen joint count (SJC); tender joint count (TJC) using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/hour]) and participant's assessment of disease activity (DA) on visual analog scale (VAS) (range 0 [very well] to 100 millimeter (mm) [extremely bad]). DAS28 less than or equal to (<=) 3.2=low DA; greater than (>) 3.2 to <=5.1=moderate DA; >5.1=high DA; <2.6=remission.
Time Frame: Month 12
Population: Full Analysis Set (FAS) included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 317
correlation coefficient | -0.06 [-0.16 to 0.06]

2. Secondary Outcome: Correlation Between Beliefs About Medicines Questionnaire Necessity Score and Safety at Month 12
Description: Correlation between BMQ necessity score and safety was assessed by using Spearman correlation coefficient. BMQ necessity: 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicate their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). Safety was assessed by analyzing the incidence, type and severity of the reported adverse events (AEs) considered related to anti-TNF- alpha therapy.
Time Frame: Month 12
Population: FAS included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 357
correlation coefficient | -0.03 [-0.13 to 0.07]

3. Secondary Outcome: Correlation Between Beliefs About Medicines Questionnaire Concerns Score and Disease Activity Score Based on 28 Joints Count at Month 12
Description: Correlation between BMQ concerns score and DAS28 score was assessed by using Pearson correlation coefficient. BMQ concerns is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Participants indicate their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). DAS28: calculated from number of SJC; TJC using 28 joints count, ESR (mm/hour) and participant's assessment of DA on VAS (range 0 [very well] to 100 mm [extremely bad]). DAS28 <=3.2= low DA; >3.2 to <=5.1= moderate DA; >5.1=high DA; <2.6=remission.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 315
correlation coefficient | 0.10 [-0.01 to 0.21]

4. Secondary Outcome: Correlation Between Beliefs About Medicines Questionnaire Concerns Score and Safety at Month 12
Description: Correlation between BMQ concerns score and safety was assessed by using Spearman correlation coefficient. BMQ Concerns is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). Safety was assessed by analyzing the incidence, type and severity of the reported AEs considered related to anti-TNF- alpha therapy.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 356
correlation coefficient | 0.03 [-0.07 to 0.13]

5. Secondary Outcome: Correlation Between Evolution of Beliefs About Medicines Questionnaire Necessity Score and Disease Activity Score Based on 28 Joints Count
Description: Correlation between evolution of BMQ necessity score and DAS28 score was assessed by calculating Pearson correlation coefficient between change from baseline in DAS28 score and BMQ necessity score at Month 6 and 12. BMQ necessity: 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicate their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). DAS28: calculated from number of SJC; TJC using 28 joints count, ESR (mm/hour) and participant's assessment of DA on VAS (range 0 [very well] to 100 mm [extremely bad]). DAS28 <=3.2= low DA; >3.2 to <=5.1= moderate DA; >5.1=high DA; <2.6=remission.
Time Frame: Month 6, 12
Population: FAS included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here, 'n' signifies those participants who were evaluable at specified time point.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
correlation coefficient
  Month 6 (n=309) | -0.05 [-0.16 to 0.06]
  Month 12 (n=285) | -0.09 [-0.20 to 0.03]

6. Secondary Outcome: Correlation Between Evolution of Beliefs About Medicines Questionnaire Necessity Score and Safety
Description: Correlation between evolution of BMQ necessity score and safety was assessed by calculating Spearman correlation coefficient between change from baseline in safety score and BMQ necessity score at Month 6 and 12. BMQ necessity: 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicate their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). Safety was assessed by analyzing the incidence, type and severity of the reported AEs considered related to anti-TNF- alpha therapy.
Time Frame: Month 6, 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
correlation coefficient
  Month 6 (n=354) | 0.01 [-0.10 to 0.11]
  Month 12 (n=334) | -0.05 [-0.16 to 0.05]

7. Secondary Outcome: Correlation Between Evolution of Beliefs About Medicines Questionnaire Concerns and Disease Activity Score Based on 28 Joints Count
Description: Correlation between evolution of BMQ concerns score and DAS28 score was assessed by calculating Pearson correlation coefficient between change from baseline in DAS28 score and BMQ concerns score at Month 6 and 12. BMQ concerns is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). DAS28: calculated from number of SJC; TJC using 28 joints count, ESR (mm/hour) and participant's assessment of DA on VAS (range 0 [very well] to 100 mm [extremely bad]). DAS28 <=3.2= low DA; >3.2 to <=5.1= moderate DA; >5.1=high DA; <2.6=remission.
Time Frame: Month 6, 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
correlation coefficient
  Month 6 (n=296) | 0.07 [-0.04 to 0.18]
  Month 12 (n=277) | 0.02 [-0.09 to 0.14]

8. Secondary Outcome: Correlation Between Evolution of Beliefs About Medicines Questionnaire Concerns and Safety
Description: Correlation between evolution of BMQ concerns score and safety was assessed by calculating Spearman correlation coefficient between change from baseline in BMQ concerns score and safety score at Month 6 and 12. BMQ concerns is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Scores obtained for individual items were summed, divided by total number of items and multiplied by 5 to give total score ranging from 5 to 25 (higher scores=stronger beliefs). Safety was assessed by analyzing the incidence, type and severity of the reported AEs considered related to anti-TNF- alpha therapy.
Time Frame: Month 6, 12
Population: FAS included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here, 'n' signifies those participants who were evaluable at each specified time point.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
correlation coefficient
  Month 6 (n=338) | 0.03 [-0.08 to 0.13]
  Month 12 (n=326) | 0.01 [-0.10 to 0.11]

9. Secondary Outcome: Percentage of Participants Agreeing or Strongly Agreeing With Beliefs About Medicines Questionnaire at Baseline
Description: BMQ consists of two 5-item scales assessing participants' agreement or strong agreement with beliefs about BMQ necessity and BMQ concerns. The items were: BMQ1: Necessity (my health at present depends on my medicines); BMQ2: Concern (having to take medications worries me); BMQ3: Necessity (my life would be impossible without my medications); BMQ4: Concern (I sometimes worry about the long term effects of my medications); BMQ5: Necessity (without my medications I would be very ill); BMQ6: Concern (my medications are mystery to me); BMQ7: Necessity (my health in the future will depend on my medications); BMQ8:Concern (my medications disrupt my life); BMQ9: Necessity (I sometimes worry about becoming too dependent on my medications); BMQ10: Concern (my medications protect me from becoming worse); BMQ11: Necessity (these medicines cause to me unpleasant adverse events).
Time Frame: Baseline
Population: BAS included all participants who were enrolled in the study and seen at baseline. Here 'n' signifies those participants who were evaluable for the given sub-scale items.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 460
percentage of participants
  BMQ1: Necessity (Agree) (n=426) | 44.6
  BMQ1: Necessity (Totally Agree) (n=426) | 49.3
  BMQ2: Concern (Agree) (n=422) | 35.5
  BMQ2: Concern (Totally Agree) (n=422) | 10.4
  BMQ3: Necessity (Agree) (n=424) | 41.3
  BMQ3: Necessity (Totally Agree) (n=424) | 43.9
  BMQ4: Concern (Agree) (n=424) | 40.6
  BMQ4: Concern (Totally Agree) (n=424) | 21.2
  BMQ5: Necessity (Agree) (n=427) | 42.9
  BMQ5: Necessity (Totally Agree) (n=427) | 37.9
  BMQ6: Concern (Agree) (n=419) | 21.0
  BMQ6: Concern (Totally Agree) (n=419) | 10.0
  BMQ7: Necessity (Agree) (n=426) | 50.2
  BMQ7: Necessity (Totally Agree) (n=426) | 38.0
  BMQ8: Concern (Agree) (n=426) | 13.4
  BMQ8: Concern (Totally Agree) (n=426) | 2.3
  BMQ9: Concern (Agree) (n=424) | 29.5
  BMQ9: Concern (Totally Agree) (n=424) | 6.8
  BMQ10: Necessity (Agree) (n=427) | 43.6
  BMQ10: Necessity (Totally Agree (n=427) | 50.8
  BMQ11: Concern (Agree) (n=428) | 16.8
  BMQ11: Concern (Totally Agree) (n=428) | 5.6

10. Secondary Outcome: Percentage of Participants Agreeing or Strongly Agreeing With Beliefs About Medicines Questionnaire at Month 6 and 12
Description: as for outcome 9
Time Frame: Month 6, 12
Population: FAS included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here 'n' signifies those participants who were evaluable at the specified time points for the given sub-scale items.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
percentage of participants
  BMQ1: Necessity (Agree)- Month 6 (n=379) | 47.0
  BMQ1: Necessity (Agree)- Month 12 (n=363) | 46.6
  BMQ1: Necessity (Totally Agree)- Month 6 (n=379) | 45.9
  BMQ1: Necessity (Totally Agree)- Month 12 (n=363) | 47.1
  BMQ2: Concern (Agree)- Month 6 (n=374) | 33.7
  BMQ2: Concern (Agree)- Month 12 (n=360) | 31.4
  BMQ2: Concern (Totally Agree)- Month 6 (n=374) | 5.3
  BMQ2: Concern (Totally Agree)- Month 12 (n=360) | 7.2
  BMQ3: Necessity (Agree)- Month 6 (n=376) | 46.0
  BMQ3: Necessity (Agree)- Month 12 (n=363) | 43.0
  BMQ3: Necessity (Totally Agree)- Month 6 (n=376) | 37.5
  BMQ3: Necessity (Totally Agree)- Month 12 (n=363) | 41.0
  BMQ4: Concern (Agree)- Month 6 (n=376) | 39.4
  BMQ4: Concern (Agree)- Month 12 (n=361) | 34.1
  BMQ4: Concern (Totally Agree)- Month 6 (n=376) | 18.6
  BMQ4: Concern (Totally Agree)- Month 12 (n=361) | 18.0
  BMQ5: Necessity (Agree)- Month 6 (n=375) | 45.3
  BMQ5: Necessity (Agree)- Month 12 (n=362) | 44.2
  BMQ5: Necessity (Totally Agree)- Month 6 (n=375) | 35.5
  BMQ5: Necessity (Totally Agree)- Month 12 (n=362) | 39.5
  BMQ6: Concern (Agree)- Month 6 (n=373) | 22.8
  BMQ6: Concern (Agree)- Month 12 (n=359) | 25.9
  BMQ6: Concern (Totally Agree)- Month 6 (n=373) | 5.9
  BMQ6: Concern (Totally Agree)- Month 12 (n=359) | 9.2
  BMQ7: Necessity (Agree)- Month 6 (n=376) | 49.2
  BMQ7: Necessity (Agree)- Month 12 (n=361) | 49.3
  BMQ7: Necessity (Totally Agree)- Month 6 (n=376) | 33.8
  BMQ7: Necessity (Totally Agree)- Month 12 (n=361) | 38.0
  BMQ8: Concern (Agree)- Month 6 (n=373) | 13.9
  BMQ8: Concern (Agree)- Month 12 (n=361) | 8.9
  BMQ8: Concern (Totally Agree)- Month 6 (n=373) | 2.4
  BMQ8: Concern (Totally Agree)- Month 12 (n=361) | 3.6
  BMQ9: Concern (Agree)- Month 6 (n=375) | 25.3
  BMQ9: Concern (Agree)- Month 12 (n=361) | 30.2
  BMQ9: Concern (Totally Agree)- Month 6 (n=375) | 6.1
  BMQ9: Concern (Totally Agree)- Month 12 (n=361) | 6.4
  BMQ10: Necessity (Agree)- Month 6 (n=380) | 51.8
  BMQ10: Necessity (Agree)- Month 12 (n=363) | 44.9
  BMQ10: Necessity (Totally Agree)- Month 6 (n=380) | 40.8
  BMQ10: Necessity (Totally Agree)- Month 12 (n=363) | 46.0
  BMQ11: Concern (Agree)- Month 6 (n=378) | 15.3
  BMQ11: Concern (Agree)- Month 12 (n=363) | 10.2
  BMQ11: Concern (Totally Agree)- Month 6 (n=378) | 5.3
  BMQ11: Concern (Totally Agree)- Month 12 (n=363) | 6.1

11. Secondary Outcome: Change From Baseline in Percentage of Participants Agreeing or Strongly Agreeing With Beliefs About Medicines Questionnaire at Month 12
Description: as for outcome 9
Time Frame: Baseline, Month 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
percentage of participants
  BMQ1: Necessity- Baseline (n=343) | 93.3
  BMQ1: Necessity- Change at Month 12 (n=343) | 0.3
  BMQ2: Concern- Baseline (n=336) | 45.8
  BMQ2: Concern-Change at Month 12 (n=336) | -7.1
  BMQ3: Necessity- Baseline (n=341) | 85.0
  BMQ3: Necessity-Change at Month 12 (n=341) | 0
  BMQ4: Concern- Baseline (n=340) | 63.5
  BMQ4: Concern-Change at Month 12 (n=340) | -11.7
  BMQ5: Necessity- Baseline (n=344) | 81.1
  BMQ5: Necessity-Change at Month 12 (n=344) | 2.9
  BMQ6: Concern- Baseline (n=339) | 30.1
  BMQ6: Concern-Change at Month 12 (n=339) | 3.5
  BMQ7: Necessity- Baseline (n=341) | 89.7
  BMQ7: Necessity-Change at Month 12 (n=341) | -2.6
  BMQ8: Concern- Baseline (n=342) | 14.0
  BMQ8: Concern-Change at Month 12 (n=342) | -1.7
  BMQ9: Concern- Baseline (n=339) | 36.3
  BMQ9: Concern-Change at Month 12 (n=339) | 0.3
  BMQ10: Necessity (n=344)- Baseline (n=344) | 94.2
  BMQ10: Necessity-Change at Month 12 (n=344) | -3.2
  BMQ11: Concern- Baseline (n=344) | 21.8
  BMQ11: Concern-Change at Month 12 (n=344) | -5.5

12. Secondary Outcome: Pearson Correlation Coefficient Between Beliefs About Medicines Questionnaire and Medication Adherence Rating Scale (MARS) at Baseline
Description: BMQ Necessity and BMQ Concerns are described in outcome measure 1 and 2 respectively. BMQ necessity-concerns: difference between necessity and concerns scales (ranges from -20 to +20, where higher score=better cost-benefit). BMQ Harm scale assesses the degree to which medicines are perceived as harmful. BMQ over use scale assesses beliefs about use of medicines and if they are overprescribed by clinicians. BMQ Harm and overuse scales comprise of 4 items, each item assessed on a 5-point scale (1=strongly disagree to 5=strongly agree). Total BMQ Harm and overuse scores were calculated as the sum of individual items and ranges from 4 to 20. Higher scores =more negative orientation towards medicines. MARS consists of a 5-item scale assessing the frequency of non-adherent behavior of participants for taking medication (5=never, 4=rarely, 3=sometimes, 2=often, 1=very often). Scores for each of the 5 items were summed; ranging from 5 to 25. Higher scores=higher levels of adherence.
Time Frame: Baseline
Population: BAS included all participants who were enrolled in the study and seen at baseline. Here, 'n' signifies those participants who were evaluable for each specified subscales.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 460
correlation coefficient
  BMQ-Necessity (n=409) | 0.13 [0.04 to 0.22]
  BMQ -Concerns (n=400) | -0.18 [-0.27 to -0.08]
  BMQ differential (Necessity-Concerns) (n=399) | 0.22 [0.12 to 0.31]
  BMQ Overuse (n=405) | -0.17 [-0.26 to -0.1]
  BMQ Harm (n=408) | -0.10 [-0.20 to -0.00]

13. Secondary Outcome: Pearson Correlation Coefficient Between Beliefs About Medicines Questionnaire and Medication Adherence Rating Scale at Month 6 and 12
Description: as for outcome 12
Time Frame: Month 6, 12
Population: FAS included all enrolled participants, who were seen at baseline and had at least 1 subsequent visit. Here, 'n' signifies those participants who were evaluable for each specified subscales.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 427
correlation coefficient
  BMQ-Necessity: Month 6 (n=366) | 0.18 [0.08 to 0.28]
  BMQ-Necessity: Month 12 (n=349) | 0.16 [0.05 to 0.26]
  BMQ -Concerns: Month 6 (n=359) | -0.15 [-0.25 to -0.05]
  BMQ -Concerns: Month 12 (n=348) | -0.24 [-0.34 to -0.14]
  BMQ (Necessity-Concerns): Month 6 (n=356) | 0.22 [0.12 to 0.31]
  BMQ (Necessity-Concerns): Month 12 (n=344) | 0.27 [0.17 to 0.37]
  BMQ Overuse: Month 6 (n=364) | -0.13 [-0.23 to -0.03]
  BMQ Overuse: Month 12 (n=349) | -0.15 [-0.26 to -0.05]
  BMQ Harm: Month 6 (n=366) | -0.11 [-0.21 to -0.00]
  BMQ Harm: Month 12 (n=350) | -0.19 [-0.29 to -0.09]

14. Secondary Outcome: Correlation Between Demographic and Clinical Factors and Beliefs About Medicines Questionnaire Necessity Score at Baseline
Description: Correlation between BMQ necessity score and participant's characteristics (demography and clinical factors) was assessed by using Pearson correlation coefficient. BMQ consists of two 5-item scales assessing participants' beliefs about necessity of prescribed medication for controlling disease (BMQ necessity) and their concerns about potential adverse consequences of taking it (BMQ concerns). Respondents indicate their degree of agreement with each statement on five-point Likert scale, ranging from 1=strongly disagree to 5=strongly agree. Total scores for necessity and concerns scales were summed; range from 5 to 25. Higher scores = stronger beliefs. Participant's characteristics included age, height, weight, body mass index (BMI), time since first RA symptoms, diagnosis, number of comorbidities and number of joint replacement or surgery.
Time Frame: Baseline
Population: BAS included all participants who were enrolled in the study and seen at baseline. Here, 'n' signifies those participants who were evaluable for the specified characteristics.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 460
correlation coefficient
  Age (n=422) | -0.030 [-0.13 to 0.07]
  Height (n=403) | -0.090 [-0.19 to 0.008]
  Weight (n=406) | -0.048 [-0.15 to 0.05]
  BMI (n=402) | -0.008 [-0.11 to 0.09]
  Time since first RA symptoms (n=409) | 0.11 [0.01 to 0.20]
  Time since first RA diagnosis (n= 422) | 0.13 [0.04 to 0.22]
  Number (No.) of comorbidities (n=422) | 0.051 [-0.04 to 0.15]
  No. of joint replacement/surgery (n= 422) | 0.053 [-0.04 to 0.15]

15. Secondary Outcome: Correlation Between Demographic and Clinical Factors and Beliefs About Medicines Questionnaire Concerns Score at Baseline
Description: Correlation between BMQ concerns score and participant's characteristics (demography and clinical factors) was assessed by using Pearson correlation coefficient. BMQ consists of two 5-item scales assessing participants' beliefs about necessity of prescribed medication for controlling disease (BMQ necessity) and their concerns about potential adverse consequences of taking it (BMQ concerns). Respondents indicate their degree of agreement with each statement on five-point Likert scale, ranging from 1=strongly disagree to 5=strongly agree. Total scores for necessity and concerns scales were summed; range from 5 to 25. Higher scores = stronger beliefs. Participant's characteristics included age, height, weight, BMI, time since first RA symptoms, diagnosis, number of comorbidities and number of joint replacement or surgery.
Time Frame: Baseline
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 460
correlation coefficient
  Age (n=409) | -0.078 [-0.17 to 0.02]
  Height (n=390) | 0.057 [-0.04 to 0.16]
  Weight (n=393) | -0.052 [-0.15 to 0.05]
  BMI (n=389) | -0.098 [-0.20 to 0.002]
  Time since first RA symptoms (n=396) | -0.06 [-0.16 to 0.04]
  Time since first RA diagnosis (n=409) | -0.08 [-0.17 to 0.02]
  No. of comorbidities (n=409) | -0.076 [-0.17 to 0.02]
  No. of joint replacement/surgery (n=409) | -0.051 [-0.15 to 0.05]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Serious Adverse Events (participants affected / at risk) | 33/460
Other Adverse Events (participants affected / at risk) | 82/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha) (N=460)
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adeocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphonia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Colon operation (Surgical and medical procedures) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 2
Osteosynthesis (Surgical and medical procedures) | 1
Peripheral endarterectomy (Surgical and medical procedures) | 1
Prolapse repair (Surgical and medical procedures) | 1
Salivary gland operation (Surgical and medical procedures) | 1
Sinus antrostomy (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Aortic stenosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha) (N=460)
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 2
Anal erosion (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Hernia (General disorders) | 1
Oedema peripheral (General disorders) | 2
Swelling (General disorders) | 1
Temperature intolerance (General disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 8
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 5
Infection (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Sinusitis aspergillus (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Viral infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Suture rupture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3
Plasma cell myelomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Morton's neuralgia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Menopausal symptom (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Bunion operation (Surgical and medical procedures) | 1
Cyst removal (Surgical and medical procedures) | 1
Ear operation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Injection (Surgical and medical procedures) | 1
Renal artery stent placement (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.